CLINICAL TRIAL: NCT01241929
Title: A Pilot Study of Using Video Images in Advance Care Planning in Patients With Advanced Cancer
Brief Title: Using Videos in Advance Care Planning for Patients With Advanced Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Angelo E. Volandes, MD, PI, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2008P000826
Record Dates: First submitted 2010-11-15; First posted 2010-11-16 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Advanced Cancer
Keywords: advanced cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- video decision aid (Experimental): Video decision aid arm
  Interventions: Behavioral: video decision aid
- Usual Care -- Verbal Description Arm (No Intervention): Verbal description of CPR (i.e., without the video).

INTERVENTIONS:
Behavioral: video decision aid — video of CPR
  Arms: video decision aid

SUMMARY:
To compare the decision making of subjects with advanced cancer having a verbal advance care planning discussion compared to subjects using a video.

DETAILED DESCRIPTION:
A.1. Aim 1: To recruit 150 subjects with advanced cancer and randomly assign these subjects to one of two advance care planning (ACP) modalities: 1. a video visually depicting CPR (intervention) or 2. a verbal narrative describing the CPR.

Hypothesis 1: It is feasible to recruit and randomize 150 subjects with advanced cancer.

A.2. Aim 2: To compare the care preferences for CPR among 150 subjects randomized to video vs. verbal narrative intervention.

Hypothesis 2: Subjects randomized to the video intervention will be significantly more likely to opt NOT to have CPR compared to those randomized to the verbal narrative.

A.3. Aim 3: To compare knowledge assessment of CPR for 150 subjects randomized to video vs. verbal narrative intervention.

Hypothesis 3: When compared to subjects randomized to the verbal narrative arm, subjects in the video group will have higher knowledge assessment scores when asked questions regarding their understanding of CPR.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of cancer that falls under one of the following: A. All patients with brain cancer, inoperable hepatocellular/bile duct/gallbladder cancer, incurable non-small cell lung carcinoma (wet IIIb or IV), extensive stage small cell lung cancer, inoperable mesothelioma, inoperable pancreatic cancer or; metastatic gastric or esophageal cancer, metastatic melanoma, OR B. Patients with the following cancers, if first-line therapy has failed and limited response is expected to second-line therapy: breast cancer, colorectal cancer, head and neck cancer, leukemia, ovarian cancer, prostate cancer, renal cancer, sarcoma, lung cancer, myeloma, or lymphoma, OR C. Less than one year prognosis.
2. ability to provide informed consent,
3. cognitive ability to participate in the study
4. ability to communicate in English.

Exclusion Criteria:

1. inability to make decisions,
2. non-English speaking,
3. new patient visit

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2009-04; Primary Completion 2012-01 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
preferences for CPR | within one hour after oncology visit
  CPR preference after visit to oncologist

SECONDARY OUTCOMES:
knowledge of CPR | baseline and post-intervention
  assess knowledge of CPR
stability of preferences | after 6-8 weeks
  assess CPR preferences again
predictors of preferences | post-intervention
  predictors of preferences for CPR

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Volandes AE, Paasche-Orlow MK, Mitchell SL, El-Jawahri A, Davis AD, Barry MJ, Hartshorn KL, Jackson VA, Gillick MR, Walker-Corkery ES, Chang Y, Lopez L, Kemeny M, Bulone L, Mann E, Misra S, Peachey M, Abbo ED, Eichler AF, Epstein AS, Noy A, Levin TT, Temel JS. Randomized controlled trial of a video decision support tool for cardiopulmonary resuscitation decision making in advanced cancer. J Clin Oncol. 2013 Jan 20;31(3):380-6. doi: 10.1200/JCO.2012.43.9570. Epub 2012 Dec 10. PMID 23233708